CLINICAL TRIAL: NCT02080065
Title: Incidence, Risk Factors, and Risk Model of Acute Kidney Injury After Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, WonHo Kim, Assistant Professor, Samsung Medical Center
Other Study IDs: 2013-12-080
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Renal Function; Liver Transplantation
Keywords: risk factor; acute kidney injury; liver transplantation; postoperative renal function
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- liver transplantation: patients who underwent living donor liver transplantation during between 2007 and 2013
  Interventions: Procedure: living donor liver transplantation

INTERVENTIONS:
Procedure: living donor liver transplantation

SUMMARY:
The incidence of acute kidney injury after liver transplantation has been reported to be 17 to 95 percent, but no definite treatment has been reported yet. Therefore, it is important to identify and prevent reversible risk factors for acute kidney injury after liver transplantation. Previous studies have reported several preoperative clinical risk factors, but preoperative medication and intraoperative colloid administration and hemodynamic parameters have not been evaluated. Therefore, we attempt to evaluate perioperative risk factors and develop simplified clinical risk scoring model.

DETAILED DESCRIPTION:
Ischemia/reperfusion injury occurs during graft harvesting, cold storage, and surgical procedures in liver transplantation. Ischemia/reperfusion injury in liver graft results in major organ damage including kidney, lung and heart as well as graft dysfunction. Graft dysfunction and renal injury after liver transplantation are major clinical issues and are associated with prognosis and low survival rate. The incidence of acute kidney injury after liver transplantation has been reported to be 17 to 95 percent, but no definite treatment has been reported yet. Therefore, it is important to identify and prevent reversible risk factors for acute kidney injury after liver transplantation. Previous studies have reported several preoperative clinical risk factors, but perioperative medication, metabolic variables (albumin, glucose, uric acid), intraoperative colloid administration and hemodynamic parameters have not been evaluated. In addition, a neutrophil-lymphocyte ratio (NLR), which has been reported to be related to systemic inflammation and associated with prognosis of cardiac and cancer patients, might be related to the development of AKI after LDLT. Therefore, we attempt to evaluate these perioperative risk factors and develop simplified clinical risk scoring model.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent living donor liver transplantation between 2010 and 2013 in Samsung Medical Center

Exclusion Criteria:

* Incomplete data regarding pre- and postoperative creatinine and estimated Glomerular Filtration Rate
* patient who underwent retransplantation

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who underwent living donor liver transplantation between 2010 and 2013
Sampling Method: Non-Probability Sample
Enrollment: 573 (Actual)
Dates: Start 2014-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
acute kidney injury as defined by RIFLE criteria | during 7 days after transplantation
  acute kidney injury as defined by RIFLE criteria

SECONDARY OUTCOMES:
incidence of renal replacement therapy | during one month after transplantation
  renal replacement therapy
incidence of acute rejection of graft | during one month after transplantation
  incidence of acute rejection of graft
incidence of initial poor graft function | during one month after transplantation
  incidence of initial poor graft function
incidence of retransplantation | during one month after transplantation
  incidence of retransplantation

OTHER OUTCOMES:
Mortality | during one month, six month, one year
  Mortality during one month, six month, one year

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea